CLINICAL TRIAL: NCT03656107
Title: The Effects of Brain Training on Brain Blood Flow: The Cognition and Flow Study
Brief Title: The Cognition and Flow Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 pandemic
Sponsor: University of Leicester (Other)
Collaborators: The Dunhill Medical Trust (Other); University Hospitals, Leicester (Other); Leicestershire Partnership NHS Trust (Other); University of Nottingham (Other); Lumosity (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0677
Record Dates: First submitted 2018-08-28; First posted 2018-09-04 (Actual); Results first posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2019-10

CONDITIONS: Dementia; Alzheimer Disease; Mild Cognitive Impairment; Aging; Cognitive Impairment
MeSH Terms: conditions — Dementia; Alzheimer Disease; Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive training (Experimental): Participants selected to brain training will be given instructions on how to access and use the program at home for 15-30minutes, 3-5 times per week for 8-12 weeks.
  Interventions: Behavioral: Cognitive Training
- Waiting-list control (No Intervention): Control participants will be waiting listed to receive the brain training program at the end of the study. control participants will undergo usual care.

INTERVENTIONS:
Behavioral: Cognitive Training — Lumosity© is a commercially available software, developed by a group of neuropsychologists, which has been used across several studies of brain training and disciplines. The brain training software targets multiple brain areas, is based online, and is relatively easy to use and administer. It has been designed to adapt to the individual's memory performance to personalise the training program to their needs. Brain exercises will be selected with the support of Lumosity© to target the following brain areas; attention, memory, visuospatial, verbal fluency, and language.
  Other Names: Brain training
  Arms: Cognitive training

SUMMARY:
About the research

There are currently 850,000 people living with dementia in the United Kingdom. It is now understand that Alzheimer's disease (AzD) can result from damaged blood vessels in the brain. Brain blood flow can be measured using ultrasound, known as transcranial Doppler ultrasonography (or TCD).

Brain training (BT) uses exercises or brain-teasers to try to make the brain work faster and more accurately. In recent years, BT has been used to try to improve memory, mood, learning, quality of life, and ability to carry out every-day activities in people with dementia.

Aims

1. To find out how acceptable and manageable this BT program is for people with dementia to undertake larger studies of BT in the future.
2. To look for any benefits for people with dementia, such as, improvements in quality of life, ability to carry out everyday tasks, mood, and brain blood flow.

How will the research be carried out?

* Forty patients with AzD, or mild cognitive impairment (MCI), and twenty healthy older adults will be recruited from memory and geriatric clinics, Join Dementia Research, general practice surgeries and community groups.
* Participants will be randomly assigned to brain training or control. The control group will be offered the program at the end of the study.
* First visit: Participants will complete questionnaires on quality of life, mood, everyday abilities, memory and an assessment of brain blood flow
* Brain training program: Participants will complete 15-30 minute sessions, 3-5 times per week
* Follow-up: participants will repeat the questionnaires and assessment of brain blood flow
* Interviews and feedback: to discuss how participants felt the program went, and find out if there are any ways it could be improved.

DETAILED DESCRIPTION:
Study design, recruitment

This will be a randomised clinical trial, undertaken at the University of Leicester, University Hospitals of Leicester (UHL) and Leicestershire Partnership National Health Service (NHS) Trusts (LPT). Following successful ethical approval, sponsorship, regulatory approvals, 40 participants with a diagnosis of MCI, or AzD, and 20 healthy volunteers will be recruited from memory clinics, general geriatric clinics, Join Dementia Research, community groups. Patients with a diagnosis of mild MCI, or mild to moderate AzD that are not under follow-up with the memory service will also be invited to participate in the study by letter invitation through their GP surgery.

Summary of the intervention

Lumosity© is a commercially available software, developed by a group of neuropsychologists, which has been used across several studies of brain training and disciplines. The brain training software targets multiple brain areas, is based online, and is relatively easy to use and administer. It has been designed to adapt to the individual's memory performance to personalise the training program to their needs. Brain exercises will be selected with the support of Lumosity© to target the following brain areas; attention, memory, visuospatial, verbal fluency, and language.

First Visit

Participants who meet the inclusion criteria, will undergo formal written consent with a member of the research team, or research delivery officer, either at home, designated LPT research space, memory service, or invited to attend the Leicester Cerebral Haemodynamics in Ageing and Stroke Medicine (CHiASM) research laboratory. Baseline assessments will be performed at this first visit including; background information on age, sex, ethnicity, medical conditions, and medication use, the Edinburgh handedness inventory (to determine left or right hand dominance), and questionnaires on mood, quality of life, and ability to carry out everyday activities. Participants who have had their baseline assessment at home will then be referred to the researcher to undertake a baseline assessment of brain blood flow at the CHiASM research space. This will be undertaken by performing selected questions from a memory test covering five major brain areas(attention, fluency, language, visuospatial and memory) with continuous TCD (ultrasound), heart rate (ECG), blood pressure (finger blood pressure monitor), and waste gases (CO2 - nasal tubes).

Randomisation

Following the collection of baseline information, participants will be chosen at random to either complete a brain training program or control. Randomisation will be performed using Sealed Envelope©. This is an online based randomisation tool which uses random permuted blocks to allocate participants to waiting list control or intervention. Participants will be enrolled and assigned a participant identification number (PIN) consecutively, and randomised to a treatment arm corresponding to the PIN. Given the nature of the trial, it is not possible to blind participants to the intervention. The Investigator will be providing weekly telephone support with the intervention, in addition to undertaking baseline and follow-up measurements, and therefore blinding of the investigator is also not possible. However, data analysis will be blinded by generating a batch anonymised data set. Randomisation will be undertaken at the initial visit. As this is an un-blinded trial, code breaking will not be required.

Intervention

Control participants will be waiting listed to receive the brain training program at the end of the study. Participants selected to brain training will be given instructions on how to access and use the program at home for 15-30minutes, 3-5 times per week for 8-12 weeks. Adherence to the program can be monitored through Lumosity©. During the 8-12 weeks participants will be provided with technical support by the investigator to minimise adherence issues and will be offered a weekly telephone call to assist with any issues that have arisen.

Follow-up

Participants will then be invited to follow up assessment at 8-12 weeks, where the TCD (ultrasound) assessment of brain blood flow will be repeated, in addition to memory testing, mood, quality of life, and ability to carry out daily activities. All travel and parking expenses to and from the study for assessments will be refunded to participants, and refreshments will be provided. No financial incentive will be offered for participating in this study. Participants will be provided with a lay summary of the results at the end of the study.

Qualitative sub-study

A qualitative study will be undertaken following the training program, which will take the form of interviews and a focus group to determine barriers and facilitators (benefits) to the brain training program. A sample of the participants who completed the brain training program and who are willing to return for interview will be included in this study. Participants will be recruited until thematic saturation is achieved (i.e. where no further themes arise from interviews or focus group). The maximum number of participants recruited to this arm would be twenty (only patient participants who have completed the intervention arm will be recruited). Where possible, the investigators will interview participants jointly with their carers in order to obtain a broader view of the impact of brain training on patients and their support network. This would allow the investigators to explore the potential wider impacts of these interventions on patients, and benefits not measured by the outcomes described above.

ELIGIBILITY:
Inclusion Criteria:

One of:

1. Healthy controls will be free of any medical co-morbidity or medication that could adversely affect cognition. Volunteers with well-controlled co-morbidities (i.e. hypertension, diabetes, will be considered for inclusion)
2. MCI as defined by National Institute on Aging and Alzheimer's Association (NIA-AA) 2011 and Petersen criteria
3. AzD as defined by the NIA-AA 2011 criteria

   And:
4. Deficits will be mild to moderate as defined by Montreal Cognitive Assessment (MoCA) score of 19-26 for MCI, and 9-18 for AzD (32-34).
5. Willing to participate
6. Capacity to consent to the study/personal consultee
7. Patients on and off anti-dementia medications will be included (acetylcholinesterase inhibitors, glutamate receptor antagonists)
8. Good understanding of written and spoken English
9. Age >50 years
10. Access to the internet and a computer/laptop or tablet device.

Exclusion Criteria:

1. Healthy controls with any medical co-morbidity or medication that could adversely affect cognition, or poorly controlled medical co-morbidities (i.e. hypertension, diabetes)
2. Unwilling to take part
3. Unable to consent/no personal consultee
4. Major medical co-morbidity; severe heart failure (ejection fraction <20%), carotid artery stenosis, severe respiratory disease, major stroke
5. Pregnancy, planning pregnancy, or lactating
6. Inadequate bilateral TCD windows
7. Participants already enrolled into other interventional studies
8. Insufficient understanding of written and spoken English
9. Age <50 years
10. No access to the internet and a computer/laptop or tablet device

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - Leicestershire Partnership Trust, Leicester, Leicestershire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beishon L, Evley R, Panerai RB, Subramaniam H, Mukaetova-Ladinska E, Robinson T, Haunton V. Effects of brain training on brain blood flow (The Cognition and Flow Study-CogFlowS): protocol for a feasibility randomised controlled trial of cognitive training in dementia. BMJ Open. 2019 May 22;9(5):e027817. doi: 10.1136/bmjopen-2018-027817. PMID 31122994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from memory services at the Leicestershire Partnership Trust, Join Dementia Research, and relatives and friends of those enrolled in the study. In addition, healthy volunteers were recruited from ongoing research studies at the University Hospitals of Leicester National Health Service Trust.
  Recruitment was from January 2019 to April 2020.
Pre-assignment Details: Participants were excluded if they did not have a temporal window for Transcranial Doppler Ultrasonography insonation. The trial was completed early due to Covid-19 and so the total number recruited (56) is less than the original planned (60).
Period: Overall Study
Arm/Group | Cognitive Training | Waiting-list Control
Started | 28 | 28
Completed | 25 | 27
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training | Waiting-list Control | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.96 (9.10) | 68.86 (8.61) | 68.41 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Successfully Recruited
Description: Feasibility
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Training | Waiting-list Control
Number analyzed (Participants) | 28 | 28
Participants | 28 | 28

2. Primary Outcome: Percentage of Participants Able to Successfully Complete the Minimum (15 Mins, 3x Per Week, for 8 Weeks) and Maximum (30 Mins, 5x Per Week, for 12 Weeks) Criteria CT Program and Complete All Assessments
Description: Feasibility
Time Frame: 17 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Training | Waiting-list Control
Number analyzed (Participants) | 28 | 28
Participants | 22 | 25

3. Primary Outcome: Percentage of Participants With Full Bilateral Data for Cerebral Blood Flow Velocity (CBFv)
Description: Feasibility CBFv as measured using transcranial Doppler ultrsonography (TCD)
Time Frame: 17 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Training | Waiting-list Control
Number analyzed (Participants) | 28 | 28
Participants | 22 | 25

4. Primary Outcome: Percentage of Control Participants Willing to be Randomised to Waiting List Control
Description: Feasibility
Time Frame: 17 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Training | Waiting-list Control
Number analyzed (Participants) | 28 | 28
Participants | 28 | 28

5. Secondary Outcome: Change in Cognition Score as Detected by the Addenbrooke's Cognitive Examination (ACE-III) From Baseline to Follow-up at 12 Weeks
Description: cognitive function. Maximum score 100, minimum score 0. Sub scale scores: attention (0-18), language (0-26), fluency (0-14), visuospatial (0-16), memory (0-26). Higher score = better cognition.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Waiting-list Control
Number analyzed (Participants) | 25 | 27
score on a scale | 0.88 (3.59) | -0.38 (3.91)

6. Secondary Outcome: Change in Functional Status - Lawton Instrumental Activities of Daily Living (IADL) From Baseline to Follow-up at 12 Weeks
Description: Functional status (maximum score =8, minimum score =0). Higher score is equivalent to better function.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Waiting-list Control
Number analyzed (Participants) | 25 | 27
units on a scale | 0.04 (0.84) | 0.04 (0.76)

7. Secondary Outcome: Change in Mood - Geriatric Depression Scale (GDS-15) From Baseline to Follow-up at 12 Weeks
Description: Mood, maximum score 15, minimum score 0. Severe depression = 10-15, mild depression = 5-9, no depression = 0-4.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Waiting-list Control
Number analyzed (Participants) | 25 | 27
units on a scale | -0.16 (1.37) | 0.41 (2.19)

8. Secondary Outcome: Change in Quality of Life Measure - Dementia Quality of Life Measure (DEMQOL) From Baseline to Follow-up at 12 Weeks
Description: Quality of life, minimum score 28, maximum score 112. higher score = better quality of life.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Waiting-list Control
Number analyzed (Participants) | 25 | 27
units on a scale | 2.12 (5.60) | -1.74 (8.66)

9. Secondary Outcome: Percentage Increase in Cerebral Blood Flow Velocity (CBFv) From Baseline to Follow-up at 12 Weeks
Description: Neurovascular function as measured by task activation, TCD protocol. Continuous CBFv was measured using TCD whilst participants underwent five cognitive tasks from the ACE-III. Task activation was measured as the percentage change in CBFv from 20 second prior to the task. T2 is the percentage change at 5-10 seconds after the task and T3 is the percentage change at 10-20 seconds after the task.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage change of CBFv
Arm/Group | Cognitive Training | Waiting-list Control
Number analyzed (Participants) | 22 | 25
percentage change of CBFv
  T2 | -1.71 (5.84) | 1.62 (5.17)
  T3 | -1.45 (4.84) | 0.39 (5.18)

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Cognitive Training | Waiting-list Control
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 3/28 | 0/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Training (N=28) | Waiting-list Control (N=28)
Drop-out (General disorders) | 3 (3) | 0 (0) — Unable to tolerate intervention resulting in drop-out from study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT03656107/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT03656107/ICF_001.pdf